CLINICAL TRIAL: NCT06931899
Title: Usefulness of Oscillometry in Assessing the Effectiveness of Inhaled Corticosteroides in Patients With COPD Exacerbator Phenotype
Brief Title: Oscillometry in the COPD Exacerbator Phenotype With Triple Inhaled Therapy Study
Acronym: OCTRIS
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other); Chiesi España, S.A.U. (Other)
Responsible Party: Principal Investigator, Yuliana Pascual González, Pneumologist, Hospital Universitari de Bellvitge
Other Study IDs: EOM018/23
Record Dates: First submitted 2025-04-03; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: Oscillometry; COPD; Inhaled corticosteroids
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Central bronchial obstruction: Oscillometry classification.
- Peripheral bronchial obstruction: Oscillometry classification.
- Pulmonary hyperinflation: Oscillometry classification.

SUMMARY:
The objective of this observational study is to determine the effectiveness of inhaled corticosteroids in patients with chronic obstructive pulmonary disease (COPD) and frequent worsening of their respiratory symptoms by using a device called an oscillometer. This instrument is capable of measuring bronchial obstruction and air trapping in the lungs through vibrations during normal breathing. The main question it seeks to answer is:

Could oscillometry be useful in assessing the effectiveness of inhaled corticosteroids in patients with COPD exacerbations, in terms of bronchial obstruction and air trapping in the lungs? Patients who choose to participate will undergo oscillometry testing and complete standard COPD questionnaires during three follow-up visits spread over three months.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is the most prevalent chronic respiratory disease worldwide, estimated at around 12% in Spain and 17.3% in Catalonia, despite significant underdiagnosis of up to approximately 74%. It is associated with high morbidity and mortality, being considered the third leading cause of death worldwide in 2021. Currently, spirometry represents the most standardized and well-known instrument for the diagnosis, control, and monitoring of COPD. However, the implementation of new tools is necessary to better define the characteristics of the disease and optimize its treatment. Furthermore, oscillometry is considered a quick and easy respiratory function test that allows the assessment of bronchial obstruction and emphysema by measuring pulmonary resistance and reactance, even in patients with normal spirometry. Its use in patients with asthma has allowed for comparisons of changes in airway obstruction with different inhaled corticosteroid (ICS) particles, with the aim of optimizing treatment choice. Therefore, its implementation in the study of patients diagnosed with COPD could also be very useful in this regard.

Main objective: To evaluate, using oscillometry, the therapeutic effectiveness of inhaled corticosteroids within triple closed therapy (LABA/LAMA/ICS) in a single device, compared to dual bronchodilation (LABA/LAMA), as maintenance treatment in patients with COPD exacerbators.

Methodology: This is an observational, prospective, multicenter study to be conducted in six hospitals in Catalonia, Spain. The goal is to include 63 patients diagnosed with COPD exacerbators, receiving dual bronchodilation treatment and meeting the endpoints for initiation of triple inhaled therapy, according to clinical practice guidelines (GesEPOC 2021, GOLD 2023). The device will be selected based on medical criteria, using the various closed-loop triple therapy inhalers currently available on the market. An initial oscillometry test will be performed to classify patients according to the predominant pattern: central obstruction, peripheral obstruction, and/or pulmonary hyperinflation. This initial measurement will be taken prior to changing treatment and immediately after the first dose of the new triple therapy inhaler. Subsequently, during patient follow-up, oscillometry will be repeated at 2, 4, and 12 weeks. The quality of life questionnaire (QLQ) and the inhaler adherence test will be self-administered at each visit. Data will be collected from the patients' electronic medical records and from laboratory tests performed during the previous year.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years.
2. Diagnosis of COPD.
3. Severe-moderate COPD measured by FEV1 and stable.
4. Patient receiving dual bronchodilation therapy (LABA/LAMA) for at least the last 4 months prior to study inclusion and meeting clinical criteria to begin triple inhaled therapy.
5. COPD exacerbations (COPD exacerbations).
6. Blood eosinophils >100 cells/mL in prior laboratory tests.
7. Patient agrees to participate in the study and signs the informed consent form.

Exclusion Criteria:

1. COPD in the last 4 weeks, with use of antibiotics or systemic corticosteroids.
2. Chronic lung disease other than COPD.
3. Severe heart failure, with frequent decompensation (in cases of mild decompensation or onset without severe heart disease, do not include the patient within 3 months of decompensation).
4. Active neoplastic processes.
5. Severe renal failure.

5. ALT greater than 2.5 times the upper limit of normal. 6. Poorly controlled insulin-dependent diabetes or involvement of 1 or more organs.

7. Positive COVID-19 test (do not include until 3 months after diagnosis by ART or COVID-19 PCR).

8. Previous treatment with ICS in the last 4 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with exacerbating COPD from the pulmonology clinics of 6 hospitals in Catalonia, Spain.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Oscillometric results | on each of the 3 visits (baseline, week 4, week 12)
  R19, R5, R5-19, X19, X5, ∆Xrs (cmH2O/(L/s)

SECONDARY OUTCOMES:
Spirometric results | initial and at visit 3 (baseline and week 12)
  FVC, FEV1
COPD Assessment Test (CAT) | on each of the 3 visits (baseline, week 4, week 12)
  score range 0-40, a higher score indicates a more severe impact of the disease on the patient's life.
Test of Adherence of Inhalers (TAI) | on each of the 3 visits (baseline, week 4, week 12)
  Items 1 to 5 assess "erratic" non-compliance (score between 5 and 25); items 6 to 10 assess "deliberate" non-compliance (score between 5 and 25); items 11 and 12 assess "unconscious" non-compliance (score between 2 and 4).
Spirometric results (forced expiratory volume in 1 second to forced vital capacity ratio) | initial and at visit 3 (baseline and week 12)
  FEV1/FVC

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Patient information can be viewed by study researchers through the REDCAP database, which has been previously coded.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: It will be available until the completion of data inclusion in the REDCAP database (approximately one year).
Access Criteria: Only the principal investigators of each center will have access to the REDCAP database.

DOCUMENTS (2):
  • Informed Consent Form: Part 1 (2023-09-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT06931899/ICF_000.pdf
  • Informed Consent Form: Part 2 (2023-09-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT06931899/ICF_001.pdf